CLINICAL TRIAL: NCT03099655
Title: Attain Stability™ Quad Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Attain Stability Quad
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Pacing; Cardiac Resynchronization Therapy; Left Ventricular Lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The Medtronic Attain Stability Quad MRI SureScan (Model 4798) is a steroid-eluting, quadripolar electrode, transvenous, over-the-wire (OTW), IS4-LLLL compatible, active fixation, cardiac vein pacing LV lead. This lead is similar to the Attain Performa family of quadripolar leads (Models 4298, 4398, and 4598) but also has a side helix for active fixation which is similar to the Attain Stability bipolar lead (Model 20066/4796) (available outside of the United States).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Attain Stability Quad Lead (Experimental): Attain Stability Quad Lead (Model 4798) - Single arm study.
  Interventions: Device: Attain Stability Quad Left Ventricular Pacing Lead

INTERVENTIONS:
Device: Attain Stability Quad Left Ventricular Pacing Lead — cardiac stimulation
  Other Names: 4798 Lead

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of the Attain Stability Quadripolar MRI SureScan Left Ventricular (LV) lead (Model 4798).

DETAILED DESCRIPTION:
The Attain Stability Quad Clinical Study is a prospective, non-randomized, multi-site, global, investigational Device Exemption (IDE), interventional clinical study. The purpose of this clinical study is to evaluate the safety and efficacy of the Attain Stability™ Quad MRI SureScan LV Lead (Model 4798). This will be assessed through a primary safety and primary efficacy endpoints.

All subjects included in the study will be implanted with a Medtronic market released de novo CRT-P or CRT-D device, compatible market released Medtronic RA and Medtronic RV leads and an Attain Stability Quad MRI SureScan LV Lead (Model 4798).

Up to 471 subjects will be enrolled into the study and up to 471 Attain Stability Quad MRI SureScan LV Lead (Model 4798) implanted, to ensure a minimum effective sample size of 400 Model 4798 leads implanted with 6 months post implant follow up visits (assuming 15% attrition) at up to 56 sites worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets CRT implant criteria as determined by local regulatory and/or hospital policy (i.e. US subjects should meet CRT device indications per the HRS/ACC/AHA guidelines)
* Patient (or legally authorized representative) has signed and dated the study-specific Informed Consent Form
* Patient is 18 years of age or older, or is of legal age to give informed consent per local and national law
* Patient is expected to remain available for follow-up visits

Exclusion Criteria:

* Patient has had a previous unsuccessful LV lead implant attempt
* Patient has a previous CRT system or LV lead implanted (for example, transvenous or epicardial)
* Patient is currently implanted with a recalled (i.e. market-withdrawn, recalled or safety alert) RA and/or RV lead
* Patient has known coronary venous vasculature that is inadequate for lead placement
* Patient has unstable angina pectoris or has had an acute myocardial infarction (MI) within the past 30 days
* Patient has had a coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past 90 days
* Patient has contraindications for standard transvenous cardiac pacing (e.g., mechanical right heart valve)
* Patient has had a heart transplant (patients waiting for heart transplants are allowed in the study)
* Patient has known renal insufficiency that would prevent them from receiving an occlusive venogram during the implant procedure
* Patient is contraindicated for <1mg dexamethasone acetate
* Patient is enrolled in any concurrent drug and/or device study that may confound the results of this study
* Patient has a terminal illness and is not expected to survive more than six months
* Patient meets exclusion criteria required by local law (e.g. age, pregnancy, breast feeding, etc.)
* Patient is unable to tolerate an urgent thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Crossley III, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (50):
- United States (35):
  - Phoenix Cardiovascular Research Group, LLC, Phoenix, Arizona
  - Sequoia Hospital, East Palo Alto, California
  - Torrance Memorial Medical Center, Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Heart Specialists Pavilion Office, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Prairie Education & Research Cooperative (Springfield IL), Springfield, Illinois
  - Iowa Heart Center (West Des Moines IA), West Des Moines, Iowa
  - Delmarva Heart Research Foundation Inc, Salisbury, Maryland
  - DLP Marquette Physicians Practices Inc, Marquette, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - HealthPartners Institute (Saint Louis Park MN), Saint Louis Park, Minnesota
  - Morristown Memorial Hospital, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Sutherland Cardiology Clinic, Memphis, Tennessee
  - Centennial Heart Cardiovascular Consultants L, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute (Plano TX), Dallas, Texas
  - CHI Saint Luke's Health - Baylor Saint Luke's Medical Center, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Kootenai Heart Clinics Northwest, Spokane, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Canada (4):
  - University of Calgary, Calgary
  - London Health Sciences Centre - University Campus, London
  - Southlake Regional Health Centre, Newmarket
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
- Germany (2):
  - Klinik für Herzchirurgie Karlsruhe, Karlsruhe
  - Berufsgenossenschaftliche Universitätsklinik Bergmannsheil GmbH, Lüdenscheid
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Azienda Ospedaliero-Universitaria Pisana - Stabilimento di Cisanello, Pisa, Italy
- Institut Jantung Negara - National Heart Institute, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Isala Zwolle, Zwolle
- Helse Bergen HF - Haukeland Universitetssjukehus, Bergen, Norway
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 471 initial enrollments;31 were excluded due to the following:
  1. No implant attempted(23)
  2. Investigator deemed not medically necessary(4)
  3. Insurance declined coverage(2)
  4. Patient did not meet criteria for the study(1)
  5. Investigator withdrew, not a good candidate(1)
  Resulting in 440 subjects with 4798 Lead implant attempted
Period: Overall Study
Arm/Group | Attain Stability Quad Lead
Started | 440
Completed | 379 (6-Month visit with original 4798 lead implanted)
Not Completed | 61

BASELINE CHARACTERISTICS:
Population: Subjects with an attempted Attain Stability Quad LV Lead implant
Groups:
- Attain Stability Quad Lead: Patients with an implant attempt for the Attain Stability Quad Lead (Model 4798)
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 329
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 312
  More than one race | 0
  Unknown or Not Reported | 73
Region of Enrollment [Number; unit: participants] — Subjects with an attempted Attain Stability Quad LV Lead implant
  participants
    Canada | 37
    Netherlands | 23
    Sweden | 3
    Hong Kong | 1
    United States | 314
    Norway | 15
    Italy | 3
    Malaysia | 23
    Germany | 12
    Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: Lead Complication-free Rate at 6 Months
Description: Subjects free of Model 4798 lead-related complications at 6 months post-implant
  -Model 4798 lead will be considered safe if the probability of subjects free from Attain Stability Quad lead-related complications at 6-months post implant is greater than 87% (i.e. the one-sided 97.5% lower confidence bound must be greater than 87%). Complications were defined in the protocol as, "An adverse event that includes the following is considered a complication: Results in death, Involves any termination of significant device function, or Requires an invasive intervention". Relationship of complication to the Attain Stability Quad lead was determined by an independent Clinical Events Committee.
Time Frame: Implant to 6 months post-implant
Population: Subjects with an attempted Attain Stability Quad Lead Model implant, results come from PMA-S Clinical Report Version 3, 28MAR2019.
Measure: Number (97.5% Confidence Interval); unit: Survival Probability (% of subjects)
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 440
Survival Probability (% of subjects) | 97.59 [96.12 to 100]

2. Primary Outcome: Proportion (Reported as a Percent) of Subjects With at Least One Vector Having PCT ≤2.5 V at 0.5 ms Pulse Width and Absence of Phrenic Nerve Stimulation (PNS)
Description: The Model 4798 LV lead has sixteen (16) programmable pacing vectors. The endpoint for the primary efficacy objective is whether or not there is at least one Model 4798 LV lead pacing vector with pacing capture voltage thresholds less than or equal to 2.5V.
  -Model 4798 lead will be considered effective if the proportion of subjects with at least one Model 4798 LV lead pacing vector with pacing capture voltage thresholds less than or equal to 2.5V at 0.5 ms pulse width (with absence of Phrenic Nerve Stimulation at 5.0 V) at 6 months post-implant is greater than 80%.
Time Frame: 6 months post-implant
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: Percent of Subjects
Groups:
- Attain Stability Quad Lead: All subjects who are successfully implanted with Model 4798 lead and with valid pacing data collected at 6 months post-implant follow-up visit.
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 377
Percent of Subjects | 96.29 [93.85 to 100]

3. Primary Outcome: Proportion (Reported as a Percent) of Subjects With at Least One Extra Vector Having PCT ≤ 4.0V at 0.5 ms Pulse Width and Absence of Phrenic Nerve Stimulation (PNS)
Description: The co-primary efficacy endpoint is whether or not a second Model 4798 lead configuration has a pacing capture threshold less than or equal to 4V, excluding the pacing vector that is already counted to the primary efficacy.
  -Model 4798 lead will be considered effective if the proportion of subjects with at least one additional Model 4798 LV lead pacing vector with pacing capture voltage thresholds less than or equal to 4.0 V at 0.5 ms pulse width (with absence of Phrenic Nerve Stimulation at 5.0 V) at 6 months post-implant is greater than 80%.
Time Frame: 6 months post-implant
Population: All subjects who are successfully implanted with a Model 4798 lead and with valid pacing data collected 6 months post-implant follow-up visit.
Measure: Number (97.5% Confidence Interval); unit: Percent of Subjects
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 377
Percent of Subjects | 94.16 [91.30 to 100]

4. Secondary Outcome: Implant Success
Description: Number of Attain Stability leads successfully implanted subjects divided by number of subjects undergo Attain Stability lead implant procedure
Time Frame: During procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 440
Percent of Subjects | 96.8 [94.7 to 98.3]

5. Secondary Outcome: Implant Duration
Description: Summary statistics including mean and standard deviation will be obtained for total implant procedure time (minutes), fluoroscopy time, and cannulation time for each successful implant procedure.
Time Frame: During procedure
Population: Subjects with a successfully implanted Attain Stability Quad Lead Model implant, results come from PMA-S Clinical Report Version 3, 28MAR2019.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Attain Stability Quad Lead: All subjects who are successfully implanted with a Model 4798 lead and with valid pacing data collected at 6 months post implant follow-up visit.
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 426
Minutes
  Implant Procedure Time | 93 (40)
  Fluoroscopy | 19 (15)
  Cannulation | 7 (11)

6. Secondary Outcome: LV Pacing Capture Threshold (PCT) at 6 Months
Description: Summary statistics including mean and standard deviation will be obtained for PCT (volt) measured at 6-month post implant visit for each successful implanted subject with valid pacing data collected at 6 months post implant follow-up visit.
Time Frame: Implant to 6 months post-implant
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 426
Volts | 1.07 (0.68)

7. Secondary Outcome: LV Impedance at 6 Months
Description: Summary statistics including mean and standard deviation will be obtained for Pacing Impedance (Ohm) measured at 6-month post implant visit for each successful implanted subject
Time Frame: Implant to 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 426
Ohms | 557.7 (179.5)

8. Secondary Outcome: Post Implant Lead Failure Rate
Description: Number of subjects with a given complication from implant through 6 months (183 days) by total number of subjects undergo Attain Stability implant procedure
Time Frame: Implant to 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Groups:
- Attain Stability Quad Lead: All subjects who are successfully implanted with a Model 4798 lead.
Arm/Group | Attain Stability Quad Lead
Number analyzed (Participants) | 426
Percent of Subjects
  Device Connection Issue | 0.23 [0.01 to 1.30]
  Device Pacing Issue | 0.23 [0.01 to 1.30]
  Device Stimulation Issue | 0.70 [0.15 to 2.20]
  Lead Dislodgement | 0.70 [0.15 to 2.20]
  Infection | 0.23 [0.01 to 1.30]
  Ventricular Tachycardia | 0.23 [0.01 to 1.30]

ADVERSE EVENTS:
Time Frame: Date of implant (or attempted implant) through study completion, an average of 6.42 months.
Arm/Group | Attain Stability Quad Lead
All-Cause Mortality (participants affected / at risk) | 22/440
Serious Adverse Events (participants affected / at risk) | 147/440
Other Adverse Events (participants affected / at risk) | 27/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attain Stability Quad Lead (N=440)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (4)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 16 (17)
Atrial flutter (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 11 (12)
Cardiac failure acute (Cardiac disorders) | 18 (21)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 15 (17)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 9 (9)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Death (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 8 (8)
Implant site pain (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Sudden cardiac death (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Pneumonia viral (Infections and infestations) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6)
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site inflammation (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Clostridium test positive (Investigations) | 1 (2)
International normalised ratio increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 4 (5)
Device connection issue (Product Issues) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 1 (1)
Device pacing issue (Product Issues) | 3 (3)
Device stimulation issue (Product Issues) | 3 (3)
Lead dislodgement (Product Issues) | 12 (12)
Oversensing (Product Issues) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 10 (11)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Medical device change (Surgical and medical procedures) | 2 (2)
Dry gangrene (Vascular disorders) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (5)
Intermittent claudication (Vascular disorders) | 2 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attain Stability Quad Lead (N=440)
Device stimulation issue (Product Issues) | 27 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03099655/SAP_000.pdf
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03099655/Prot_001.pdf